CLINICAL TRIAL: NCT01536106
Title: Intracoronary Infusion of Concentrated Autologous Bone Marrow Mononuclear Cells in Acute Myocardial Infarction Patients Utilizing a Novel Point-of-Care Device for Rapid-Delivery of Stem Cells (AMIRST)
Brief Title: Rapid Delivery of Autologous Bone Marrow Derived Stem Cells in Acute Myocardial Infarction Patients.
Acronym: AMIRST
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: TotipotentRX Cell Therapy Pvt. Ltd. (Industry)
Collaborators: TotipotentRX Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TPRX/POC/BMSC/AMIRST/1.0
Record Dates: First submitted 2011-07-16; First posted 2012-02-20 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Acute Myocardial Infarction
Keywords: Cell therapy, Bone marrow stem cells, cardiac cell therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Implantation of bone marrow derived mononuclear cells
  Interventions: Other: Autologous Bone marrow mononuclear cells
- Placebo Control (Placebo Comparator): Infusion of autologous peripheral blood
  Interventions: Other: Placebo control

INTERVENTIONS:
Other: Autologous Bone marrow mononuclear cells — Intracoronary administration of concentrated BMMNC on the same day of BM aspiration using point of care technology.
  Other Names: BMMNC treatment group
  Arms: Treatment
Other: Placebo control — Intracoronary infusion of autologous peripheral blood.
  Other Names: Placebo control group
  Arms: Placebo Control

SUMMARY:
The primary objective of the study is to determine the feasibility and safety of intracoronary administration of autologous bone marrow derived mononuclear cell product in patients at risk for clinically significant cardiac dysfunction following AMI.

The secondary objective of the study is to assess the effect on cardiac function and infarct region perfusion. A concurrent placebo control patient group meeting eligibility but not receiving autologous bone marrow derived stem cells will be evaluated similar to the treated group to assess the rate of significant spontaneous improvement in cardiac function.

DETAILED DESCRIPTION:
Emerging evidence indicate that progenitor stem cells derived from bone marrow can be used to improve cardiac function in acute myocardial infarction patients. There is a great potential for stem cell therapy, using a variety of cell precursors to contribute to new blood vessel formation and muscle preservation in the myocardial infarct zone. The administration of cells via an infusion through the infarct related artery appears to be feasible and result in a clinical effect in some studies. Across the globe AMI is the leading cause of morbidity and mortality. This cannot be prevented by optimal standard therapies i.e. balloon or stent dilation of the infarct vessels.

The study is a double blind, placebo controlled, randomized, multicenter trial. Male or female patients between 18-75 years with first incidence of Acute Myocardial Infarction(AMI) and LVEF less than or equal to 40% are included in the study. Patients who have undergone successful percutaneous intervention (PCI) within ≤ 24 hours after onset of symptoms (PTCA/stent) or / and Thrombolysed patients having TIMI-3 flow are eligible to take part in the study.

A total of 30 subjects will be recruited and randomly assigned to receive concentrated BMMNC or placebo. All patients will undergo bone marrow aspiration within 3-10 days from the index event(infarction). Bone Marrow(BM) will be processed utilizing point of care technology. Following cell processing, the concentrated BMMNC or placebo control is infused directly into the infarct related artery using the stop flow method. Clinical follow up for all the subjects at 1,30, 60, 90, 180 and 360 days will be performed from the day of the procedure, with primary and secondary end points evaluated for both study arms.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female of age 18 - 75 years
* Incidence of first myocardial infarction
* Acute STEMI with LV hypokinesia involving anteroseptal, lateral or inferior walls
* LVEF < 40% pre-intervention
* Successful percutaneous intervention (PCI) within ≤ 24 hours after onset of symptoms (PTCA/stent) or / and Thrombolysed patients having TIMI-3 flow.
* Written informed consent

Exclusion Criteria:

* Multi-vessel coronary disease requiring surgical intervention (CABG) or left main coronary artery disease > 50% blockage
* Previous history of CABG
* Pulmonary edema
* Cardiogenic shock
* Myocarditis
* Renal or hepatic dysfunction
* Hematologic disease

General Exclusion Criteria:

* Alcohol or drug dependency, active or uncontrolled acute myocarditis
* HIV, HBV, or HCV infections
* Evidence of malignant or hematological diseases
* Metal implants of any kind
* Claustrophobia
* Renal insufficiency
* History of bleeding disorder
* Anemia (haemoglobin <8.5mg/dl)
* Platelet count <100,000/ml

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-01 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events as a measure of safety | 12 Months
  Feasibility and safety of Intracoronary infusion of autologous BMMNCs processed through intraoperative point of care technology, freedom from arrhythmia's.

SECONDARY OUTCOMES:
Changes in the global Left Ventricular Ejection Fraction(LVEF), LV volumes-End Systolic Volume (ESV) and End Diastolic Volume (EDV), infarct size, myocardial mass, myocardial viability and regional wall motion abnormalities. | 12 Months
  Changes in the global Left Ventricular Ejection Fraction(LVEF), LV volumes-End Systolic Volume (ESV) and End Diastolic Volume (EDV), infarct size, myocardial mass, myocardial viability and regional wall motion abnormalities measured by Cardiac MRI and assessed by central Core lab.
Major adverse cardiac events (MACE) | 12 Months
  MACE was defined as the composites of any cause of death, myocardial infarction, revascularization of the target vessel, re-hospitalization for heart failure, and life-threatening arrhythmia.
Quality of life | 12 Months
  Quality of life assessment is done using short-form 36, Minnesota living with heart failure questionnaire and Seattle Angina Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Venkatesh Ponemone, PhD, Study Director — TotipotentRX Cell Therapy Pvt. Ltd.; Kenneth Harris, MS, Study Chair — TotipotentRX Cell Therapy Pvt. Ltd.; Ashok Seth, FRCP, FACC, Principal Investigator — Fortis Escorts Heart Institute and Research Centre; Upendra Kaul, MD,DM, FACC, Principal Investigator — Fortis Flt. Lt. Rajan Dhall Hospital; Sreenivas A Kumar, MD, DM, FACC, Principal Investigator — CARE Hospitals Hyderabad, India
Locations (3):
- India (3):
  - CARE Hospitals, Banjara Hills, Hyderabad, Hyderabad
  - Fortis Escorts Heart Institute and Research Centre, New Delhi, New Delhi
  - Fortis Flt. Lt. Rajan Dhall Hospital, New Delhi, New Delhi

REFERENCES:
- [Result] Roncalli J, Mouquet F, Piot C, Trochu JN, Le Corvoisier P, Neuder Y, Le Tourneau T, Agostini D, Gaxotte V, Sportouch C, Galinier M, Crochet D, Teiger E, Richard MJ, Polge AS, Beregi JP, Manrique A, Carrie D, Susen S, Klein B, Parini A, Lamirault G, Croisille P, Rouard H, Bourin P, Nguyen JM, Delasalle B, Vanzetto G, Van Belle E, Lemarchand P. Intracoronary autologous mononucleated bone marrow cell infusion for acute myocardial infarction: results of the randomized multicenter BONAMI trial. Eur Heart J. 2011 Jul;32(14):1748-57. doi: 10.1093/eurheartj/ehq455. Epub 2010 Dec 2. PMID 21127322
- [Result] Strauer BE, Yousef M, Schannwell CM. The acute and long-term effects of intracoronary Stem cell Transplantation in 191 patients with chronic heARt failure: the STAR-heart study. Eur J Heart Fail. 2010 Jul;12(7):721-9. doi: 10.1093/eurjhf/hfq095. PMID 20576835
- [Result] Dohmann HF, Silva SA, Sousa AL, Braga AM, Branco RV, Haddad AF, Oliveira MA, Moreira RC, Tuche FA, Peixoto CM, Tura BR, Borojevic R, Ribeiro JP, Nicolau JC, Nobrega AC, Carvalho AC. Multicenter double blind trial of autologous bone marrow mononuclear cell transplantation through intracoronary injection post acute myocardium infarction - MiHeart/AMI study. Trials. 2008 Jul 3;9:41. doi: 10.1186/1745-6215-9-41. PMID 18598362